CLINICAL TRIAL: NCT01270737
Title: A Double-blind Randomized Controlled Trial on Whole Soy and Daidzein Supplementation on Reduction of Blood Pressure in Prehypertensive Postmenopausal Chinese Women
Brief Title: Whole Soy and Daidzein on Reduction of Blood Pressure in Postmenopausal Chinese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Prof. Suzanne C Ho, director of Center of Research and Promotion of Women's Health, CRPWH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CUHKGRF465810
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2010-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — daidzein; Refit milk powder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whole soy (Active Comparator)
  Interventions: Dietary Supplement: Whole soy (soy flour)
- daidzein (Active Comparator)
  Interventions: Dietary Supplement: daidzein
- milk powder (Placebo Comparator)
  Interventions: Dietary Supplement: milk powder

INTERVENTIONS:
Dietary Supplement: Whole soy (soy flour) — 40g soy flour per day for six months
  Other Names: soy flour
  Arms: Whole soy
Dietary Supplement: daidzein — 66mg daidzein per day for six months
  Arms: daidzein
Dietary Supplement: milk powder — 40g low-fat dry milk per day for six months
  Other Names: dry milk
  Arms: milk powder

SUMMARY:
The investigators hypothesize that whole soy or purified daidzein alone could reduce blood pressure and CVD risks in equol-producing menopausal Chinese women.

DETAILED DESCRIPTION:
Hypertension is an important risk factor for cardiovascular diseases. Substantial evidence has also shown that prehypertension [systolic blood pressure (BP) 120-139 mm Hg or diastolic BP 80-89 mm Hg] is the strongest predictor of incident hypertension and is associated with elevated risk of cardiovascular diseases. Thus, prehypertension and its progression to hypertension have enormous public health implications. Soybean contains many beneficial components, among which isoflavones have received most research attention. Recently researchers have investigated their influences on vascular functions but only a handful of studies have focused on BP reduction as the primary outcome.The role of whole soy or daidzein on BP is yet unclear.

The investigators hypothesize that whole soy (soy flour) or purified daidzein alone could reduce BP,and decrease CVD risks in menopausal women with prehypertension or initial untreated hypertension. The investigators propose to perform a 24-week double-blind, randomized, placebo-controlled trial in postmenopausal women with prehypertension or stage 1 hypertension. The primary objective is to verify if whole soy (soy flour) or purified daidzein alone has anti-hypertensive effects at a dosage of habitual high soy intake.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Chinese women with prehypertension or stage 1 hypertension

Exclusion Criteria:

* Medical treatment for blood pressure or lipids reduction hormones replacement therapy in recent 3 months, chronic renal or hepatic diseases

Ages: 48 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
24 hours blood pressure | 1 year
  24 hour ambulatory blood pressure recording

SECONDARY OUTCOMES:
Cardiovascular Disease (CVD) risks | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C Ho, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Center of Research and Promotion of Women's Health, Hong Kong, China

REFERENCES:
- [Derived] Liu ZM, Chen B, Li S, Li G, Zhang D, Ho SC, Chen YM, Ma J, Qi H, Ling WH. Effect of whole soy and isoflavones daidzein on bone turnover and inflammatory markers: a 6-month double-blind, randomized controlled trial in Chinese postmenopausal women who are equol producers. Ther Adv Endocrinol Metab. 2020 Jun 18;11:2042018820920555. doi: 10.1177/2042018820920555. eCollection 2020. PMID 32595918
- [Derived] Liu ZM, Li G, Zhang D, Ho SC, Chen YM, Ma J, Huang Q, Li S, Ling WH. Effect of whole soy and purified daidzein on androgenic hormones in chinese equol-producing post-menopausal women: a six-month randomised, double-blinded and Placebo-Controlled trial. Int J Food Sci Nutr. 2020 Aug;71(5):644-652. doi: 10.1080/09637486.2020.1712682. Epub 2020 Jan 9. PMID 31914834
- [Derived] Liu ZM, Ho SC, Chen YM, Tomlinson B, Ho S, To K, Woo J. Effect of whole soy and purified daidzein on ambulatory blood pressure and endothelial function--a 6-month double-blind, randomized controlled trial among Chinese postmenopausal women with prehypertension. Eur J Clin Nutr. 2015 Oct;69(10):1161-8. doi: 10.1038/ejcn.2015.24. Epub 2015 Mar 18. PMID 25782428
- [Derived] Liu ZM, Ho SC, Chen YM, Tang N, Woo J. Effect of whole soy and purified isoflavone daidzein on renal function--a 6-month randomized controlled trial in equol-producing postmenopausal women with prehypertension. Clin Biochem. 2014 Sep;47(13-14):1250-6. doi: 10.1016/j.clinbiochem.2014.05.054. Epub 2014 May 27. PMID 24877660
- [Derived] Liu ZM, Ho CS, Chen YM, Woo J. Can soy intake affect serum uric acid level? Pooled analysis from two 6-month randomized controlled trials among Chinese postmenopausal women with prediabetes or prehypertension. Eur J Nutr. 2015 Feb;54(1):51-8. doi: 10.1007/s00394-014-0684-1. PMID 24659208
- [Derived] Liu ZM, Ho SC, Chen YM, Ho S, To K, Tomlinson B, Woo J. Whole soy, but not purified daidzein, had a favorable effect on improvement of cardiovascular risks: a 6-month randomized, double-blind, and placebo-controlled trial in equol-producing postmenopausal women. Mol Nutr Food Res. 2014 Apr;58(4):709-17. doi: 10.1002/mnfr.201300499. Epub 2013 Nov 24. PMID 24273218
- [Derived] Liu ZM, Ho SC, Woo J, Chen YM, Wong C. Randomized controlled trial of whole soy and isoflavone daidzein on menopausal symptoms in equol-producing Chinese postmenopausal women. Menopause. 2014 Jun;21(6):653-60. doi: 10.1097/GME.0000000000000102. PMID 24149925
- [Derived] Liu ZM, Ho SC, Chen YM, Woo J. A six-month randomized controlled trial of whole soy and isoflavones daidzein on body composition in equol-producing postmenopausal women with prehypertension. J Obes. 2013;2013:359763. doi: 10.1155/2013/359763. Epub 2013 Aug 1. PMID 23984051